CLINICAL TRIAL: NCT05085951
Title: Randomised Controlled Trial (Feasibility Study) of Prophylactic Pyloric Balloon Dilatation During Ivor Lewis Oesophagectomy to Prevent Delayed Gastric Emptying
Brief Title: Prophylactic Pyloric Balloon Dilatation During Ivor Lewis Oesophagectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 21/SUR/574
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Postprocedural Delayed Gastric Emptying

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic pyloric balloon dilatation (Experimental): OGD and dilatation
  Interventions: Device: 20 mm CRE balloon
- No endoscopic intervention (Placebo Comparator): OGD but no dilatation
  Interventions: Diagnostic Test: OGD

INTERVENTIONS:
Device: 20 mm CRE balloon — Endoscopic balloon that is used to dilate pylorus
  Arms: Prophylactic pyloric balloon dilatation
Diagnostic Test: OGD — OGD (No dilatation)
  Arms: No endoscopic intervention

SUMMARY:
This is a feasibility study to assess recruitment for a randomised control trial comparing prophylactic pyloric ballon dilatation versus control group (no intervention) in Ivor-Lewis Oesophagectomy

DETAILED DESCRIPTION:
The Ivor Lewis gastro-oesophagectomy is a complex operation that is performed to treat cancer of the oesophagus (food pipe) whereby most of the oesophagus and upper stomach are removed and the remaining stomach is brought into the chest and joined to the remaining oesophagus. In order to reduce the burden of complications of the procedure, research has been conducted in search of methods to improve the procedure and outcomes after the operation. Delayed gastric emptying (how quickly food empties out of your stomach into your small bowel) is a common problem after this operation (20% of patients). The situation can lead to a feeling of being full up, loss of appetite and nausea. Rarely, in severe cases patients may vomit or food going into lung causing a chest infection or develop a leak from the operative joint which can prolong hospital stay by an average of 5 days. Treatment currently is uncertain, as is the scale of problem (how common it is) and there is no standard definition for delayed gastric emptying (there is no agreed standard way to describe slow emptying of food from the stomach into the small bowel by experts). There is a theory that the problem might be caused due to the outlet of the stomach (pylorus) narrowing down. Prevention of the problem is also uncertain.

In order to investigate prevention of the problem, the study will involve randomising patients during the oesophagectomy to either dilatation (stretching) of the pylorus with a balloon, or not, and completion of an abbreviated quality of life questionnaire (8 multiple choice questions).

During the oesophagectomy, all patients routinely have endoscopy (camera test of the gullet and stomach) to assess the tumour. It is during this part of the operation that you will be randomised to either the balloon group or no intervention. The questionnaire is to assess your quality of life, in terms of delayed gastric emptying, at different points after the operation.

Preoperative endoscopic pyloric balloon dilatation with 20 mm has been shown to decrease incidence of DGE (only 18.3 % of the intervention group developed DGE compared to 37.5% in the non-intervention group (Hadzijusufovic et al., 2019). This however was a cohort study, and the main issue was that the intervention group had 115 patients whilst the non-dilatation group had 24 patients (tumour could not be passed with the scope). There aren't currently any published randomised control trials that looked at intra-operative endoscopic pyloric dilatation and how this relates to incidence of DGE.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 undergoing Ivor Lewis oesophagectomy in Derriford.

Exclusion Criteria

* Patient declined to participate.
* Impassable stricture at endoscopy.
* Patient is unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of delayed gastric emptying | less than 14 days post op
  Chest X-ray and Nasogastric tube output

SECONDARY OUTCOMES:
Rate of anastomotic leak | less than 14 days post op
  If clinical indication diagnosis will be with CT
Rate of pneumonia | less than 14 days post op
  If clinically indicated by CXR or CT

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Rollinson, Study Chair — University Hospitals Plymouth NHS Trust
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No